CLINICAL TRIAL: NCT00858689
Title: Add-on Pilot Trial of Minocycline in Fragile X Syndrome
Brief Title: Add-on Pilot Trial of Minocycline to Treat Fragile X Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FRAXA Research Foundation (Other)
Collaborators: Fragile X Research Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010308
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Fragile X Syndrome
Keywords: Clinical Drug Trial
MeSH Terms: conditions — Fragile X Syndrome | interventions — Minocycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- minocyline 50 mg or 100 mg PO BID (Experimental): open label treatment with minocycline low or high dose, 50 mg or 100 mg PO (by mouth) BID (twice a day), added to existing medication regimen for 8 weeks
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — 50-100 mg PO BID for 8 weeks with an option for a 1 year extension.
  Other Names: Solodyn, Dynacin, Arestin, Minocin

SUMMARY:
Fragile X Syndrome (FXS) is the most common known inherited form of mental impairment, developmental disability and autism. Minocycline is an antibiotic that has recently been used to treat the mouse model for Fragile X, and was found to reverse the structural abnormalities that are seen their brain cells. The purpose of this research study is to determine if minocycline is an effective treatment for patients with fragile X syndrome (FXS).

DETAILED DESCRIPTION:
Fragile X Syndrome (FXS) is the most common known inherited form of mental impairment and is also associated with a range of learning disabilities, neurological problems, such as seizures, and behavioural difficulties. For many individuals with FXS, behavioral difficulties result in severe problems within the family and community, particularly in the form of agitation, temper outbursts, hyperactivity, and aggression. These problems often require a variety of psychopharmacological and behavioural approaches. Although a variety of medications can be helpful in FXS there are no targeted interventions based on molecular abnormalities that have been studied. Defects in dendritic spine formation have been found in the brains of patients with Fragile X, suggesting these structures may represent an anatomical and physiological basis for the cognitive deficits associated with this disorder. Recent research has suggested that minocycline may have a specific benefit in the treatment of FXS. Minocycline is an antibiotic that has been found to inhibit the activity of matrix metallo-proteinase-9 (MMP-9), which is up-regulated in the hippocampus of FMR1 KO (Fragile X Mental Retardation-1 Knockout) mice and may be responsible for the immature dendritic spine profile of hippocampal neurons. Minocycline has recently been used to treat the FXS KO mouse model for Fragile X, and was found to rescue this abnormal phenotype by inducing the formation of mature dendritic spines in FMR1 KO hippocampal neurons, both in vitro and in vivo. Minocycline treated FXS KO mice also performed significantly better in the elevated maze, a cognitive performance test that measures activity and anxiety.

Exciting preclinical effects of minocycline with regard to the FXS disease model have led to this pilot proposal, which is designed to generate preliminary data that could be used to support a larger clinical trial.

The overall hypothesis is that minocycline is a specific molecular targeted treatment for FXS that will display beneficial effects on disruptive behaviour and possibly other associated features of FXS via a reduction in MMP-9 activity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FXS by clinical evaluation and confirmed by FMR1-DNA testing with presence of full mutation or mosaicism for the full mutation. Prior DNA testing reports will be accepted, when available.
* Age between 13 to 35 years inclusive at the time of informed consent.
* Male or female
* CGI-Severity Score of 4 or greater, indicative of moderate or greater severity of behavioural problems. This is a 7-point scale of clinical global impression of severity that the clinician fills out after considering all the available information on the patient, including the parent history, the examination in clinic, reports from the school and other sources.
* Score of 9 or greater on the Aberrant Behaviour Checklist - Irritability Scale (top 50th %-tile). The ABC is a global behaviour checklist implemented for the measurement of drug and other treatment effects in mentally impaired individuals. It is made up of 5 empirically derived dimensions including irritability, lethargy/withdrawal, inappropriate speech, hyperactivity, and stereotypic behaviour based on 58 items that describe various behavioural problems.
* Availability of parent and/or caregiver for all clinic visits and assessments.
* English language fluency and reading level of 6th grade or greater in one caregiver.

Exclusion Criteria:

* Allergy to minocycline.
* Kidney disease or elevated renal function tests.
* Liver disease or elevated liver function tests.
* Participants with neutropenia, anemia, or thrombocytopenia.
* History of systemic lupus erythematosus or screening anti-nuclear antibody (ANA) titre of >1:40, as minocycline may cause a lupus-like reaction.
* Individuals who do not have a mother or caregiver who is willing to participate in the clinic visits.
* Individuals who are pregnant or at risk to become pregnant, specifically sexually active females will be excluded.
* Presence of persistent psychotic symptoms
* Subjects with symptom severity likely judged to endanger personal safety or safety of others.
* History of systemic lupus erythematosus or screening anti-nuclear antibody (ANA) titre of >1:40, as minocycline may cause a lupus-like reaction.

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2007-10; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Paribello, M.D., Principal Investigator — Fragile X Research Foundation of Canada
Locations (1):
- Surrey Place Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Paribello C, Tao L, Folino A, Berry-Kravis E, Tranfaglia M, Ethell IM, Ethell DW. Open-label add-on treatment trial of minocycline in fragile X syndrome. BMC Neurol. 2010 Oct 11;10:91. doi: 10.1186/1471-2377-10-91. PMID 20937127
- See also: The Fragile X Research Foundation of Canada is a non-profit organization which is dedicated to funding biomedical research for improved treatment and, ultimately, a cure for fragile X. — http://www.fragile-x.ca
- See also: FRAXA is a non-profit organization whose mission is to accelerate progress toward effective treatments and a cure for Fragile X, by funding the most promising research. — http://www.fraxa.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty subjects with FXS between 13 and 35 years of age were enrolled between December 2007 and June 2008, and after baseline testing they were started on an 8-week treatment course of minocycline added on to any other medications being administered at the time of enrollment.
Pre-assignment Details: Inclusion criteria included (1) diagnosis of FXS by clinical evaluation and confirmed by FMR1-DNA testing with presence of full mutation or mosaicism for the full mutation.
Groups:
- Minocyline 50 mg or 100 mg PO BID: open label, single arm study of minocyline 50 mg or 100 mg PO BID
Period: Overall Study
Arm/Group | Minocyline 50 mg or 100 mg PO BID
Started | 20
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Minocyline 50 mg or 100 mg PO BID: open label minocyline 50 mg or 100 mg PO BID
Arm/Group | Minocyline 50 mg or 100 mg PO BID
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 9
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Region of Enrollment [Number; unit: participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline of ABC Irritability Subtest Score at 8 Weeks
Description: The 15-item Irritability Scale includes questions about aggression, self-injury, tantrums, agitation, and unstable mood on a scale of 0 to 45 with higher scores indicating greater severity. This scale has been successfully used in previous medication studies in children with autism and in patients with FXS and in a controlled trial of ampakine CX516 in FXS. All ABC subscales showed good reliability when used by parents and caregivers of individuals with FXS to assess behavior in the CX516 study NCT00054730, and yielded intraclass correlation coefficient (ICC) values of 0.7-0.9.
Time Frame: Baseline and 8 weeks
Population: ABC-I change in subjects completing 8 weeks of minocycline treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocyline 50 mg or 100 mg PO BID
Number analyzed (Participants) | 19
units on a scale | -14.37 (7.84)

2. Primary Outcome: ABC Irritability Subtest Score
Description: ABC Irritability subtest score was used
Time Frame: 8 weeks
Population: completed 8 weeks of minocycline treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Minocyline 50 mg or 100 mg PO BID
Number analyzed (Participants) | 19
units on a scale | 7.74 (4.82)

3. Primary Outcome: ABC Irritability Subtest Score
Description: ABC (Aberrant behavior checklist) Irritability subtest score was used
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: Parent Defined Target Symptoms Scale-Visual
Time Frame: Baseline
Reporting Status: Not Posted

5. Secondary Outcome: Clinical Global Impression Scale
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Stanford Binet 5 (SB5)
Time Frame: Baseline
Reporting Status: Not Posted

7. Secondary Outcome: The Peabody Picture Vocabulary Test Third Edition (PPVT-III)
Time Frame: Baseline
Reporting Status: Not Posted

8. Secondary Outcome: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Time Frame: Baseline
Reporting Status: Not Posted

9. Secondary Outcome: Non-Verbal Associative Learning Task (NVALT)
Time Frame: Baseline
Reporting Status: Not Posted

10. Secondary Outcome: Vineland Adaptive Behaviour Scales (VABS)
Time Frame: Baseline
Reporting Status: Not Posted

11. Secondary Outcome: Parent Defined Target Symptoms Scale-Visual
Time Frame: 8 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Parent Defined Target Symptoms Scale-Visual
Time Frame: 1 year
Reporting Status: Not Posted

13. Secondary Outcome: Clinical Global Impression Scale
Time Frame: 8 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Clinical Global Impression Scale
Time Frame: 1 year
Reporting Status: Not Posted

15. Secondary Outcome: Stanford Binet 5 (SB5)
Time Frame: 1 year
Reporting Status: Not Posted

16. Secondary Outcome: The Peabody Picture Vocabulary Test Third Edition (PPVT-III)
Time Frame: 8 weeks
Reporting Status: Not Posted

17. Secondary Outcome: The Peabody Picture Vocabulary Test Third Edition (PPVT-III)
Time Frame: 1 year
Reporting Status: Not Posted

18. Secondary Outcome: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Time Frame: 8 weeks
Reporting Status: Not Posted

19. Secondary Outcome: The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Time Frame: 1 year
Reporting Status: Not Posted

20. Secondary Outcome: Non-Verbal Associative Learning Task (NVALT)
Time Frame: 8 weeks
Reporting Status: Not Posted

21. Secondary Outcome: Non-Verbal Associative Learning Task (NVALT)
Time Frame: 1 year
Reporting Status: Not Posted

22. Secondary Outcome: Vineland Adaptive Behaviour Scales (VABS)
Time Frame: 8 weeks
Reporting Status: Not Posted

23. Secondary Outcome: Vineland Adaptive Behaviour Scales (VABS)
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Minocyline 50 mg or 100 mg PO BID
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minocyline 50 mg or 100 mg PO BID (N=20)
Increased serum ANA titre (Immune system disorders) | 2 (2) — two participants developed an asymptomatic seroconversion of their ANA, both exhibiting a 1/80 titre with a nucleolar pattern

LIMITATIONS AND CAVEATS:
This was an open-label trial. Further study in a randomized controlled trial is warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No